CLINICAL TRIAL: NCT04423016
Title: Clinical Determinants of Cerebrovascular Reactivity in Very Preterm Infants During the Transitional Period
Brief Title: Transitional Cerebrovascular Reactivity in Very Preterm Infants
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: NEO-TOHRx
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Cerebral Autoregulation; Preterm Birth; Premature Infant Disease
Keywords: cerebral autoregulation; cerebrovascular reactivity; preterm infants; transitional period
MeSH Terms: conditions — Premature Birth | interventions — Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Near Infrared Spectroscopy monitoring — Non-invasive continuous monitoring of cerebral oxygenation
Device: Electrical velocimetry and pulse oximetry — Non-invasive continuous monitoring of cerebral oxygenation

SUMMARY:
The transitional period, defined as the first 72 hours after preterm birth, is often characterized by a significant hemodynamic instability and may also be associated with an impairment of cerebral autoregulation, with relevant clinical implications. The moving correlation coefficient between cerebral oxygenation and heart rate, also defined as TOHRx, has been previously proposed as a marker of cerebrovascular reactivity and provides an indirect estimation of cerebral autoregulation in preterm infants.

This study aims to evaluate whether different antenatal, perinatal and postnatal factors may influence cerebrovascular reactivity in very preterm infants during the transitional period.

DETAILED DESCRIPTION:
The transitional period, defined as the first 72 hours after preterm birth, is often characterized by a significant hemodynamic instability and may also be associated with an impairment of cerebral autoregulation, with relevant clinical implications. The moving correlation coefficient between cerebral oxygenation and heart rate, also defined as TOHRx, has been previously proposed as a marker of cerebrovascular reactivity and provides an indirect estimation of cerebral autoregulation in preterm infants.

This prospective observational study aims to evaluate whether different antenatal, perinatal, and postnatal factors may influence cerebrovascular reactivity in very preterm infants during the transitional period.

Infants <32 weeks' gestation are enrolled within 12h from birth. A simultaneous monitoring of cerebral oxygenation (CrSO2) by near-infrared spectroscopy and of heart rate (HR) by pulse oximetry and electrical velocimetry is performed continuously over the first 72h.

The moving correlation coefficient between CrSO2 and HR is calculated using the ICM+ software (Cambridge Enterprise Ltd) using 5-min, 30-point epochs. Time periods with evidence of major artefacts, or with a missing data proportion >50% are excluded from this calculation. Positive TOHRx values will be interpreted as markers of impaired autoregulation.

A screening echocardiogram is routinely performed at the time of enrollment and repeated 6-12 hourly in the presence of a patent ductus arteriosus (PDA) or 12-24 hourly if there is no evidence of PDA. Based on echocardiographic features, the ductal status is classified as follows: no evidence of PDA, restrictive PDA (restrictive shunt pattern and left atrium to aortic root ratio [LA:Ao] ratio <1.5), hemodynamically significant PDA (pulsatile shunt pattern, LA:Ao ratio ≥1.5 or presence of reversed end-diastolic flow either in the descending aorta or in the anterior cerebral artery).

A concomitant cerebral ultrasound scan, aimed at evaluating brain parenchyma and the occurrence of prematurity-related complications, such as intraventricular hemorrhage, is also performed.

During the study period, the following antenatal and neonatal data are tracked down on a specific case report form: gestational age (GA); birth weight (BW); non-invasive blood pressure; antenatal steroids (complete course vs. incomplete course or not given); evidence of reversed end-diastolic flow at antenatal umbilical Doppler (uREDF) (present vs. absent); ventilatory status over the first 72 hours of life (mechanical ventilation, continuous positive airway pressure [CPAP], nasal cannulas or self-ventilating in air [SVIA]); surfactant administration; development of IVH over the first 72 hours of life; ongoing inotropes (dopamine, dobutamine or both).

The correlation between antenatal, perinatal, and postnatal clinical variables and TOHRx is going to be evaluated using generalized linear mixed models or generalized estimating equations.

ELIGIBILITY:
Inclusion Criteria:

* gestational age <32 weeks' gestation

Exclusion Criteria:

* major congenital malformations
* congenital heart disease

Ages: 1 Day to 3 Days | Sex: All
Age Groups: Child
Study Population: Preterm infants <32 weeks' gestation during the transitional period (0-72 hours of life)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
Correlation between TOHRx and gestational age | 0-72 hours
  Correlation between TOHRx and gestational age
Correlation between TOHRx and antenatal steroids administration | 0-72 hours
  Correlation between TOHRx and antenatal steroids administration (full course vs. incomplete course or not given)
Correlation between TOHRx and antenatal Doppler status | 0-72 hours
  Correlation between TOHRx and antenatal Doppler status (normal or abnormal)
Correlation between TOHRx and ductal status | 0-72 hours
  Correlation between TOHRx and ductal status (hemodynamically significant, restrictive or closed)
Correlation between TOHRx and respiratory support | 0-72 hours
  Correlation between TOHRx and respiratory support modality (mechanical ventilation, CPAP, nasal cannulas or self-ventilating in air)
Correlation between TOHRx and inotropes | 0-72 hours
  Correlation between TOHRx and inotropes administration (dopamine; dobutamine; dopamine and dobutamine)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Corvaglia, MD, Principal Investigator — S. Orsola-Malpighi University Hospital, Bologna, Italy
Locations (1):
- Sant'Orsola-Malpighi University Hospital, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No